CLINICAL TRIAL: NCT02164565
Title: The Use of Tranexamic Acid (TXA) Intravenously, to Reduce Blood Loss in Proximal Femur Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104-12-EMC
Record Dates: First submitted 2014-05-29; First posted 2014-06-16 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Femur Surgery
MeSH Terms: interventions — Tranexamic Acid; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (TXA) treatment (Experimental): Tranexamic Acid (TXA) treatment
  Interventions: Drug: Tranexamic Acid (TXA) treatment
- control grup: without Tranexamic Acid (TXA) treatment. (Experimental): control grup: without Tranexamic Acid (TXA) treatment.
  Interventions: Drug: control grup: without Tranexamic Acid (TXA) treatment.

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) treatment — Tranexamic Acid (TXA) treatment
  Arms: Tranexamic Acid (TXA) treatment
Drug: control grup: without Tranexamic Acid (TXA) treatment. — control grup: without Tranexamic Acid (TXA) treatment.
  Arms: control grup: without Tranexamic Acid (TXA) treatment.

SUMMARY:
The use of Tranexamic Acid (TXA) intravenously, to Reduce Blood Loss in proximal femur surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60, who came to the orthopedic department for proximal femur fracture surgery
* Sound judgment

Exclusion Criteria:

* Known hypersensitivity to Tranexamic Acid or component solution provided
* Subarachnoid hemorrhage
* Acquired color blindness
* Myocardial infarction in 12 months before admission
* Unstable angina
* Known clotting disorders (Thromboembolic disease in the past, elongated PT and PTT, hypercoagulability),
* Kidney or liver failure
* Another situation prostate resection , pathologic fractures according to anamnesis or by imaging
* Oncology patients
* Patients on anticoagulation
* Patients undergoing vascular intervention ( coronary or peripheral ), which was inserted Supporter requires a Dual antiplatelet therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of blood loss in ml. | up to 13 months
  Hbloss=BV X (Hbi - Hbe) X 0.001 + Hbt Hbi - hemoglobin level before the surgery ) gram X liter-1(. Hbe - hemoglobin level 3 days after the surgery ( gram X liter-1). Hbt - The amount of hemoglobin that was given in the blood transfusion (gram). Hbloss - Change of hemoglobin loss.
  After calculating the amount of loss of hemoglobin, the volume of blood lost can be found:
  Blood loss = 1000 X Hbloss/ Hbi
  Evaluation of blood loss will be through:
  1. Comparing hemoglobin level before and after surgery and calculation of quantitative Change of hemoglobin loss.
  2 .Registration evaluating blood loss at the end of surgery 3. Collecting and recording blood drain. 4. Tracking Blood Transfusion. Of course we collect the data: assessment of bleeding in the analysis, the number of blood units given, the amount of blood collected drain

CONTACTS AND LOCATIONS:
Overall Officials: Nimrod Rozen, Prof., Principal Investigator — Division of Orthopedic & Rehabilitatio, HaEmek Medical Center
Locations (1):
- Orthopedic Department, HaEmek Medical Center, Afula, Israel